CLINICAL TRIAL: NCT06501768
Title: A Pilot Clinical Trial of Cardiovascular Genistein Therapy for Heart Failure Inflammation
Brief Title: Cardiovascular Genistein Therapy for Heart Failure Inflammation
Acronym: CARDIOGEN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Greenstone Biosciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARDIOGEN
Record Dates: First submitted 2024-07-01; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genistein Therapy (Experimental): Participants will consume 250 mg of genistein BID (500 mg total) by mouth for the first 4 weeks before blood samples are collected. And then, patients will take 500 mg of genistein BID (1000 mg total) for the next 4 weeks before blood are collected. Afterward, patients will take 750 mg of genistein BID (1500 mg total) for 4 weeks before blood samples are collected. Afterward, patients will be off Genistein for 6 weeks before returning for blood sample collection. The Genistein capsules are manufactured and obtained from MCS Formulas. The genistein is certified to be 98% pure genistein by HPLC and is good laboratory practice (GLP) certified. At baseline, and again before Genistein discontinuation (at 12 weeks), we will also perform transthoracic echocardiography and a 6-minute walk test.
  Interventions: Drug: Genistein

INTERVENTIONS:
Drug: Genistein — Escalation genistein dosing, followed by wash-out period

SUMMARY:
This Phase 1b/2a open-label study is designed to assess the safety and efficacy of genistein in patients with heart failure (HF). The investigation will focus on its impact on inflammatory and cardiometabolic biomarkers, as well as its effects on cardiac function and exercise capacity.

Blood samples will be collected at baseline, following each administration of genistein, and after a six-week placebo washout period. These samples will be subjected to comprehensive analyses to evaluate inflammatory cytokines and novel molecular markers. Routine tests, including Complete Blood Count (CBC), Basic Metabolic Panel (Chem 7), Liver Function Tests (LFT), Hemoglobin A1c (HbA1c), N-terminal pro b-type natriuretic peptide (NT-proBNP), C-Reactive Protein (CRP), and troponin T will be performed. Advanced assessments will include RNA sequencing (RNA-seq) on peripheral blood mononuclear cells (PBMCs) and the isolation of plasma exosomes to identify inflammatory biomarkers. In addition, a subset of the blood samples will be used to generate induced pluripotent stem cells (iPSCs) to further explore the treatment's impact on heart failure-related inflammatory markers.

Echocardiography, in accordance with the European Society of Cardiology (ESC) and the American Heart Association (AHA) guidelines, will be utilized to evaluate cardiac structure and function with a specific focus on the left and right ventricular functions and valvular integrity. Exercise capacity will be gauged through a standardized six-minute walk test. Levels of NT-proBNP will be measured as an indicator of cardiac stress and function.

Participants will be followed up for 18 weeks post-enrolment, with the primary endpoint being the change in inflammatory markers from baseline to the three-month mark. Secondary endpoints will include changes in cardiac function and exercise capacity over the same period. The trial aims to enrol 40 participants, following ethical committee approval and the acquisition of written informed consent. Each patient will receive genistein at a dosing regimen starting with 250 mg twice daily (BID) for 4 weeks, escalating to 500 mg BID for the subsequent 4 weeks, and 750 mg BID for another 4 weeks, culminating in a 6-week follow-up period.

The insights garnered from this study are expected to be pivotal in guiding future larger-scale studies and to elucidate the therapeutic potential of genistein in the management of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of heart failure of ischemic or nonischemic etiology with LVEF <40%.
* ATTR cardiomyopathy with any LVEF.
* Stable optimally tolerated dosages of HF therapies for 3 months with no change in medical management regimen for at least 1 month.
* NT-proBNP >350 pg/mL.

Exclusion Criteria:

* Coronary intervention in the past 3 months.
* Pregnancy
* Cancer
* Patients on a vegan diet
* Patients taking supplements such as isoflavonoid or resveratrol.
* Ethanol abuse (men: >4 drinks on any day or more than 14 drinks by week; women: >3 drinks on any day or more than 7 drinks per week)
* Liver dysfunction (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3X ULN or total bilirubin greater than 1.5 times ULN)
* Renal dysfunction (eGFR less than 25 mL/min/1.73 m2)
* Uncontrolled diabetes (HgbA1c >10%)
* Coagulopathies
* Cytopenia (leukocytopenia or hemoglobin < 9 mg/dl or platelets <100x103/mm3)
* Any patients who had been hospitalized in the past 3 months for reasons other than heart failure.
* NYHA Functional Class I or Functional Class IV symptoms.
* Acute bacterial or viral infectious disease, or acute exacerbation of a chronic infectious disease
* Known hypersensitivity to soy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
HF inflammatory and cardiometabolic markers | 18 weeks
  To comprehensively assess the safety profile and determine the impact of Genistein on key inflammatory and cardiometabolic biomarkers in patients with HF, the following markers will be assessed using specific measurement tools:
  Inflammatory Markers:
  * Interleukin-6 (IL-6): Measured using ELISA.
  * Interleukin-8 (IL-8): Measured using ELISA.
  * Tumor Necrosis Factor-alpha (TNF-α): Measured using ELISA.
  * Interferon-gamma (IFN-γ): Measured using ELISA.
  Cardiometabolic Markers:
  * B-type Natriuretic Peptide (BNP): Measured using immunoassay.
  * C-reactive Protein (CRP): Measured using immunoassay.
  * Hemoglobin A1C (HgA1C): Measured using standard laboratory methods.
  * Complete Blood Count (CBC): Measured using automated hematology analyzer.
  * Comprehensive Metabolic Panel (Chem 7): Measured using standard laboratory methods.
  * Liver Function Tests (LFT): Measured using standard laboratory methods.

SECONDARY OUTCOMES:
Exercise capacity and cardiac performance | 18 weeks
  Exercise capacity will be evaluated by 6-minute walk test, which will be performed by a blinded observer according to the standard protocol.
  Cardiac performance will be evaluated by echocardiography. The scans will assess left ventricle end-systolic- and end-diastolic volumes (LVESV and LVEDV), myocardial mass, assessment of LV systolic and diastolic function, left ventricular ejection fraction (LVEF), radial and longitudinal global- and segmental strain by two-dimensional speckle-tracking echocardiography (2D-STE), LV diastolic function will be assessed by E lateral and medial velocity, E/e', LA volume, and TR velocity). A comprehensive assessment of RV size, RV systolic and diastolic function, RV systolic pressures, RV 2D speckle tracking derived longitudinal strain analysis of the RV free wall averaged over three segments of the RV free wall (2D-STE), assessment of the valvular function and tissue Doppler parameters (e', s') will be performed.

OTHER OUTCOMES:
Blood biomarkers | 18 weeks
  We will aim to examine alterations in blood biomarkers through unbiased proteomics using the SEER or OLink platform post-Genistein treatment and benchmark against baseline. The specific biomarkers and measurement tools are as follows:
  Proteomics Analysis:
  * Platform: OLink or RayBiotech proteomic profiling array.
  * Biomarkers: A comprehensive panel of proteins related to inflammation, oxidative stress, and cardiovascular health will be assessed.
  * Examples of Biomarkers:
    * Cytokines: IL-6, IL-8, TNF-α, IFN-γ.
    * Acute Phase Proteins: CRP, Serum Amyloid A.
    * Growth Factors: VEGF, EGF.
    * Metabolic Proteins: Adiponectin, Leptin.
  Units of Measure:
  • The biomarkers will be measured in their respective units, typically in picograms per milliliter (pg/mL) or nanograms per milliliter (ng/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No